CLINICAL TRIAL: NCT04662320
Title: Promoting Healing of Nerves Through Electrical Stimulation
Acronym: PHONES
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Checkpoint Surgical Inc. (Industry)
Collaborators: Congressionally Directed Medical Research Programs (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0153-CSP-001; W81XWH1920065 (Other Grant/Funding Number: Department of Defense USAMRAA)
Record Dates: First submitted 2020-11-24; First posted 2020-12-10 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Cubital Tunnel Syndrome; Nerve Compression; Nerve Injury; Ulnar Neuropathies
Keywords: Therapeutic Electrical Stimulation; Nerve Regeneration; Nerve Healing; Nerve Injury; Cubital Tunnel; Ulnar Nerve
MeSH Terms: conditions — Cubital Tunnel Syndrome; Neuroma; Ulnar Neuropathies | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Brief Electrical Stimulation (Experimental): Single, 10 minute dose of electrical stimulation delivered to the ulnar nerve during surgical intervention for cubital tunnel decompression.
  Interventions: Device: Checkpoint BEST System
- Standard of Care (No Intervention): Surgical intervention for cubital tunnel decompression.

INTERVENTIONS:
Device: Checkpoint BEST System — Single use medical device, consisting of electric stimulator and intraoperative lead. Therapy consists of single, 10 minute dose delivered proximal to site of decompression/repair.
  Other Name: Checkpoint BEST System
  Other Names: Brief Electrical Stimulation (BES) Therapy
  Arms: Brief Electrical Stimulation

SUMMARY:
This study is evaluating a new therapeutic use of electrical stimulation to promote nerve healing and improve functional recovery following surgical intervention for nerve compression. A single dose of the therapeutic stimulation is delivered as part of the surgical intervention to address compression of the ulnar nerve at the elbow.

DETAILED DESCRIPTION:
Preliminary research has shown that delivering a brief period of electrical stimulation following nerve repair promotes nerve healing and functional recovery. This study is investigating the use of a single dose of therapeutic electrical stimulation to promote nerve healing. The therapy is delivered as part of the surgical intervention to address compression of the ulnar nerve at the elbow, commonly referred to as Cubital Tunnel Syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Electrodiagnostic evidence of ulnar neuropathy at the elbow.
* Are candidates for surgical intervention.
* Evidence of motor involvement such as intrinsic muscle atrophy or weakness.
* Are age 18-80 years.
* Signed and dated informed consent form.

Exclusion Criteria:

* Severe comorbid condition, such as arrythmia or congestive heart failure, preventing surgery
* Previous history or current transection of ulnar nerve, or concomitant upper extremity nerve injury
* Global peripheral neuropathy affecting the hands
* Age less than 18 or greater than 80 years
* Un-affected hand maximum grip strength <12kg

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change in Grip Strength at 1 year. | 1 year
  Change in grip strength at 1 year from baseline (pre-operative) assessment.

SECONDARY OUTCOMES:
Grip Strength | Pre-surgery, 6 weeks, 3 months, 5 months, 7 months, 9 months, and 1 year
  Maximum grip strength
Lateral Pinch Strength | Pre-surgery, 6 weeks, 3 months, 5 months, 7 months, 9 months, and 1 year
  Maximum lateral pinch strength
2-point discrimination | Pre-surgery, 6 weeks, 3 months, 5 months, 7 months, 9 months, and 1 year
  Evaluation of sensory function, measuring tactile discrimination.
Semmes-Weinstein Monofilament Testing | Pre-surgery, 6 weeks, 3 months, 5 months, 7 months, 9 months, and 1 year
  Evaluation of sensory function, measuring pressure detection threshold.
Medical Research Council (MRC) motor grading. | Pre-surgery, 6 weeks, 3 months, 5 months, 7 months, 9 months, and 1 year
  Grading of muscle strength on 0 to 5 scale, with higher score representing greater function.
Maximal finger spread measurement. | Pre-surgery, 6 weeks, 3 months, 5 months, 7 months, 9 months, and 1 year
  Measurement of maximal finger spread.
Patient Reported Outcome Measurement System (PROMIS) Upper Extremity Function | Pre-surgery, 10 days, 6 weeks, 3 months, 5 months, 7 months, 9 months, and 1 year
  Questionnaire providing patient reported estimate of upper extremity function on a 0-100 scale with >50 representing greater normal function.
Patient Reported Outcome Measurement System (PROMIS) Pain Interference | Pre-surgery, 10 days, 6 weeks, 3 months, 5 months, 7 months, 9 months, and 1 year
  Questionnaire providing patient reported estimate of interference of pain on daily activities on a 0-100 scale with >50 representing greater than normal pain interference on daily activities.
Michigan Hand Questionnaire (MHQ) | Pre-surgery, 10 days, 6 weeks, 3 months, 5 months, 7 months, 9 months, and 1 year
  MHQ is a patient reported estimate of hand function on a 0-100 scale with a higher number indication greater hand function.
Nerve Conduction Velocity (NCV) | Pre-surgery, 3 months, and 7 months
  Measurement of how quickly an electrical impulse moves along the nerve.
Electromyography (EMG) | Pre-surgery, 3 months, and 7 months
  Measurement of the electrical activity in a muscle.

CONTACTS AND LOCATIONS:
Overall Officials: Amy M Moore, MD, Principal Investigator — The Ohio State Univeristy Department of Plastic and Reconstructive Surgery
Locations (5):
- United States (5):
  - Stanford University, Stanford, California
  - Northwestern Feinberg School of Medicine - Department of Orthopaedic Surgery, Chicago, Illinois
  - Washington University in St. Louis, St Louis, Missouri
  - The Ohio State Univeristy - Department of Plastic and Reconstructive Surgery, Columbus, Ohio
  - Medical College of Wisconsin - Hand Center, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Saffari TM, Walker ER, Pet MA, Moore AM. Brief Intraoperative Electrical Stimulation to Enhance Nerve Regeneration. Plast Reconstr Surg Glob Open. 2024 Apr 10;12(4):e5730. doi: 10.1097/GOX.0000000000005730. eCollection 2024 Apr. No abstract available. PMID 38600968
- [Background] Power HA, Morhart MJ, Olson JL, Chan KM. Postsurgical Electrical Stimulation Enhances Recovery Following Surgery for Severe Cubital Tunnel Syndrome: A Double-Blind Randomized Controlled Trial. Neurosurgery. 2020 Jun 1;86(6):769-777. doi: 10.1093/neuros/nyz322. PMID 31432080
- [Background] Gordon T, Amirjani N, Edwards DC, Chan KM. Brief post-surgical electrical stimulation accelerates axon regeneration and muscle reinnervation without affecting the functional measures in carpal tunnel syndrome patients. Exp Neurol. 2010 May;223(1):192-202. doi: 10.1016/j.expneurol.2009.09.020. Epub 2009 Oct 1. PMID 19800329
- [Background] Jo S, Pan D, Halevi AE, Roh J, Schellhardt L, Hunter Ra DA, Snyder-Warwick AK, Moore AM, Mackinnon SE, Wood MD. Comparing electrical stimulation and tacrolimus (FK506) to enhance treating nerve injuries. Muscle Nerve. 2019 Nov;60(5):629-636. doi: 10.1002/mus.26659. Epub 2019 Aug 21. PMID 31397919
- [Background] Evans A, Padovano WM, Patterson JMM, Wood MD, Fongsri W, Kennedy CR, Mackinnon SE. Beyond the Cubital Tunnel: Use of Adjunctive Procedures in the Management of Cubital Tunnel Syndrome. Hand (N Y). 2023 Mar;18(2):203-213. doi: 10.1177/1558944721998022. Epub 2021 Apr 2. PMID 33794683
- [Background] Sayanagi J, Acevedo-Cintron JA, Pan D, Schellhardt L, Hunter DA, Snyder-Warwick AK, Mackinnon SE, Wood MD. Brief Electrical Stimulation Accelerates Axon Regeneration and Promotes Recovery Following Nerve Transection and Repair in Mice. J Bone Joint Surg Am. 2021 Oct 20;103(20):e80. doi: 10.2106/JBJS.20.01965. PMID 34668879
- [Background] Roh J, Schellhardt L, Keane GC, Hunter DA, Moore AM, Snyder-Warwick AK, Mackinnon SE, Wood MD. Short-Duration, Pulsatile, Electrical Stimulation Therapy Accelerates Axon Regeneration and Recovery following Tibial Nerve Injury and Repair in Rats. Plast Reconstr Surg. 2022 Apr 1;149(4):681e-690e. doi: 10.1097/PRS.0000000000008924. PMID 35139047